CLINICAL TRIAL: NCT05490355
Title: Radiofrequency Ablation and Steroid Versus Steroid Alone for Relief of Pain in Patients With Advanced Knee and Hip Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ended prematurely due to low enrollment interest.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Avneesh Chhabra, Chief, Musculoskeletal Radiology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0337
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Osteoarthritis; perineural steroid injections; radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineural Steroid Injections Alone (Active Comparator): Participants assigned to this study arm will receive only Perineural Steroid Injections per clinical standards.
  Participant will also complete a joint function questionnaire at 4 time points, pre-procedure, 2 weeks post procedure, 3 months post procedure, and 6 months post procedure.
  Interventions: Procedure: Perineural Steroid Injection
- Perineural Steroid Injections Plus Radiofrequency Ablation (Experimental): Participants assigned to this study arm will receive Perineural Steroid Injections plus Radiofrequency Ablation per clinical standards.
  Participant will also complete a joint function questionnaire at 4 time points, pre-procedure, 2 weeks post procedure, 3 months post procedure, and 6 months post procedure.
  Interventions: Procedure: Radiofrequency Ablation (RFA); Procedure: Perineural Steroid Injection

INTERVENTIONS:
Procedure: Radiofrequency Ablation (RFA) — RFA involves heating of periarticular nerves using continuous RFA (80-90C for 60-90 seconds) that results in electromodulation and denervation reducing pain. It can be done under fluoroscopy or CT guidance. CT guidance has additional benefit of better localization of the nerves, as opposed to simple bony landmarks used in fluoroscopy, since nerve branching variations are common and will be used in this study.
  Arms: Perineural Steroid Injections Plus Radiofrequency Ablation
Procedure: Perineural Steroid Injection — Perineural Steroid Injections involve CT guided injection of Local Anesthetic and Steroid into a nerve root of the spine to provide ongoing pain relief.

SUMMARY:
The purpose of this trial is to determine if radiofrequency ablation plus steroid perineural injections at the knee or hip provide longer pain relief and better function to patients than the current standard of care, perineural steroid injections alone.

This pilot study is a prospective two arm randomized trail, all participants will be recruited from the University of Texas Southwestern Medical Center (UTSW) outpatient orthopedic clinic. 40 participants (20 hip and 20 knee OA) will be enrolled into the standard of care arm (treated with steroid injections alone) and 40 participants (20 hip and 20 knee OA) will be enrolled into the investigational arm (treatment with a combination of radiofrequency ablation (RFA) plus steroid injections) for a total of 80 enrolled participants. All subjects will complete a function and pain assessment at the time of injection and three additional time points: 2 weeks, 3 months, and 6 months post injection. This study will use the same knee function questionnaire and frequency currently used in clinic per standard of care. In addition, all participant's surgical history and prior injection history will be reviewed via the Electronic Medical Record (EMR).

ELIGIBILITY:
Inclusion Criteria: (1 & 2 or 3)

1. Males or females age 18 to 100 years
2. Osteoarthritis of the knee Kellgren-Lawrence grade 3-4 OR
3. Osteoarthritis of the hip Tonnis grades 2 or higher

Exclusion Criteria:

1. History of knee or hip replacement
2. History of intra-articular steroid injections within the past 6 weeks
3. Active infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Hip Functional score at baseline (pre-procedure) | Baseline (Pre-Procedure)
  Hip functional score will be assessed using current standard of care Hip score questionnaire for hip OA at baseline (pre-procedure). Possible scores range from 1-100, where lower scores indicate worse function.
Hip Functional score at 2 weeks post procedure | 2 weeks post procedure
  Hip functional score will be assessed using current standard of care Hip score questionnaire for hip OA at 2 weeks post procedure. Possible scores range from 1-100, where lower scores indicate worse function.
Hip Functional score at 3 months post procedure | 3 months post procedure
  Hip functional score will be assessed using current standard of care Hip score questionnaire for hip OA at 3 months post procedure. Possible scores range from 1-100, where lower scores indicate worse function.
Hip Functional score at 6 months post procedure | 6 months post procedure
  Hip functional score will be assessed using current standard of care Hip score questionnaire for hip OA at 6 months post procedure. Possible scores range from 1-100, where lower scores indicate worse function.
Knee Functional score as measured by standard of care questionnaire for knee OA at baseline (pre-procedure) | Baseline (pre-procedure)
  Knee functional score will be measured using current standard of care questionnaire for knee osteoarthritis (OA) at baseline (pre-procedure). Possible scores range from 1-100, where higher scores indicate worse function.
Knee Functional score as measured by standard of care questionnaire for knee OA at 2 weeks post procedure | 2 weeks post procedure
  Knee functional score will be measured using current standard of care questionnaire for knee osteoarthritis (OA) at 2 weeks post procedure. Possible scores range from 1-100, where higher scores indicate worse function.
Knee Functional score as measured by standard of care questionnaire for knee OA at 3 months post procedure | 3 months post procedure
  Knee functional score will be measured using current standard of care questionnaire for knee osteoarthritis (OA) at 3 months post procedure. Possible scores range from 1-100, where higher scores indicate worse function.
Knee Functional score as measured by standard of care questionnaire for knee OA at 6 months post procedure | 6 months post procedure
  Knee functional score will be measured using current standard of care questionnaire for knee osteoarthritis (OA) at 6 months post procedure. Possible scores range from 1-100, where higher scores indicate worse function.

CONTACTS AND LOCATIONS:
Overall Officials: Avneesh Chhabra, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen AF, Mullen K, Casambre F, Visvabharathy V, Brown GA. Thermal Nerve Radiofrequency Ablation for the Nonsurgical Treatment of Knee Osteoarthritis: A Systematic Literature Review. J Am Acad Orthop Surg. 2021 May 1;29(9):387-396. doi: 10.5435/JAAOS-D-20-00522. PMID 32701684
- [Background] Conger A, McCormick ZL, Henrie AM. Pes Anserine Tendon Injury Resulting from Cooled Radiofrequency Ablation of the Inferior Medial Genicular Nerve. PM R. 2019 Nov;11(11):1244-1247. doi: 10.1002/pmrj.12155. Epub 2019 May 24. No abstract available. PMID 30859692
- [Background] Kim SY, Le PU, Kosharskyy B, Kaye AD, Shaparin N, Downie SA. Is Genicular Nerve Radiofrequency Ablation Safe? A Literature Review and Anatomical Study. Pain Physician. 2016 Jul;19(5):E697-705. PMID 27389113
- [Background] Li G, Zhang Y, Tian L, Pan J. Radiofrequency ablation reduces pain for knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2021 Jul;91:105951. doi: 10.1016/j.ijsu.2021.105951. Epub 2021 Apr 18. PMID 33882358
- [Background] Rivera F, Mariconda C, Annaratone G. Percutaneous radiofrequency denervation in patients with contraindications for total hip arthroplasty. Orthopedics. 2012 Mar 7;35(3):e302-5. doi: 10.3928/01477447-20120222-19. PMID 22385437
- [Background] Chye CL, Liang CL, Lu K, Chen YW, Liliang PC. Pulsed radiofrequency treatment of articular branches of femoral and obturator nerves for chronic hip pain. Clin Interv Aging. 2015 Mar 16;10:569-74. doi: 10.2147/CIA.S79961. eCollection 2015. PMID 25834413
- [Background] Bhatia A, Hoydonckx Y, Peng P, Cohen SP. Radiofrequency Procedures to Relieve Chronic Hip Pain: An Evidence-Based Narrative Review. Reg Anesth Pain Med. 2018 Jan;43(1):72-83. doi: 10.1097/AAP.0000000000000694. PMID 29140960